CLINICAL TRIAL: NCT06469957
Title: Impact of Hospital Pharmacist on Drug Management in Patients With Bronchopulmonary Cancer Treated by Chemotherapy and/or Immunotherapy or Oral Targeted Therapy
Brief Title: Impact of Hospital Pharmacist on Drug Management in Patients With Bronchopulmonary Cancer
Acronym: IMPACTO
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2023-12
Record Dates: First submitted 2024-06-03; First posted 2024-06-24 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Patients With Bronchopulmonary Cancer
Keywords: Hospital pharmacist; Pharmaceutical intervention; Chemotherapy / Immunotherapy /oral targeted therapy; Bronchopulmonary cancer
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires and data collection sheet — Questionnaires

SUMMARY:
This is a prospective, non-interventional study to evaluate impact of hospital pharmacist on drug management in patients (only questionnaires) with bronchopulmonary cancer treated by Chemotherapy and/or Immunotherapy or Oral targeted therapy. The primary objective of the study is to evaluate the number of unscheduled consultations/hospitalizations during 6 months.

DETAILED DESCRIPTION:
Currently, several treatments can be used for bronchopulmonary cancers: targeted oral therapy (OCT), oral chemotherapy, iv chemotherapy, iv immunotherapy. These therapies are rather unknown to community pharmacy and induce several adverse effects and drug interactions. These treatments require collaboration between different professionals (community and hospital pharmacists) in order to allow follow up and security in patient supportive care.

In our context of shortage of care staff, with a polymedicated and elderly population, we would like to assess the impact of hospital pharmacist in the drug management for patient with bronchopulmonary cancers treated by these therapies.

Other French studies (Lille, Angers, Tours) involving hospital pharmacists were carried out and aimed to evaluate the number of pharmaceutical interventions carried out without assessing the impact on the patient. In addition, no study concerns the Center Val de Loire region.

The aim of the study is to impact of hospital pharmacist (interview) on the number of unscheduled consultations/hospitalizations.

This is a prospective, non-interventional study to evaluate impact of hospital pharmacist on drug management in patients with bronchopulmonary cancer. Participants will be included after being informed and after obtaining no opposition to participate. Data collection sheet will be performed by hospital pharmacist at inclusion. Participants will be treated according to standard of care for cancer treatment. An interview will be performed 1 month, 3 months and 6 months after inclusion between hospital pharmacist and participant to obtain information's on cancer treatments (questionnaires). These interviews will be performed by phone or when the patient comes to the hospital for a follow-up consultation as part of the treatment of his cancer (standard of care).

A total of 60 participants will be included in this study based on 1) the number of patients received a novel cancer treatment in the center during 12 months and 2) considered eligibility criteria, pharmacist availability and patients consent.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years
2. Patient without cognitive impairments
3. Patient with bronchopulmonary cancer
4. Patient treated by chemotherapy, immunotherapy or oral targeted therapy

Exclusion Criteria:

1. Patient informed and opposed to participate
2. Language barrier and lack of translator
3. Patient under guardianship, curatorship or deprived of liberty
4. Pregnant or breastfeeding women
5. Participation in any drug clinical drug trials
6. Patient with no insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bronchopulmonary cancer who received a new treatment with oral targeted therapy, chemotherapy or immunotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-12-27 (Estimated)

PRIMARY OUTCOMES:
Impact of hospital pharmacist (interview) on the number of unscheduled consultations/hospitalizations. | From enrolment to the end of the follow up phase (6 months)
  Number of unscheduled consultations or hospitalizations during the follow up phase

SECONDARY OUTCOMES:
Impact of hospital pharmacist (interview) on cancelled consultations/hospitalizations rate | From enrolment to the end of the follow up phase (6 months)
  Number of cancelled consultations/hospitalizations
Impact of hospital pharmacist (interview) on treatment observance (number of dispensation) | From enrolment to the end of the follow up phase (6 months)
  Number of treatment dispensation
Impact of hospital pharmacist (interview) on treatment observance (gap between dispensation) | From enrolment to the end of the follow up phase (6 months)
  Gap between each treatment dispensation
Impact of hospital pharmacist (interview) on adverse effects | From enrolment to the end of the follow up phase (6 months)
  Number of adverse effects (follow up phase of 6 months)
Impact of hospital pharmacist (interview) on adverse effects leading to interrupted or withdrawn treatment | From enrolment to the end of the follow up phase (6 months)
  Number of adverse effects leading to interrupted or withdrawn treatment
Impact of hospital pharmacist on pharmaceutical intervention | From enrolment to the end of the follow up phase (6 months)
  Number of pharmaceutical interventions (eg. inappropriate prescription, drug interactions)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine DA VIOLANTE, Dr, Principal Investigator — CHU d'Orléans
Locations (1):
- CHU d'Orléans, Orléans, France

REFERENCES:
- [Background] Babin M, Folliard C, Robert J, Sorrieul J, Kieffer H, Augereau P, Devys C. [Pharmaceutical consultations in oncology: Implementation, one-year review and outlooks]. Ann Pharm Fr. 2019 Sep;77(5):426-434. doi: 10.1016/j.pharma.2019.05.001. Epub 2019 Jul 7. French. PMID 31288930